CLINICAL TRIAL: NCT05858905
Title: Forward-Shifted Intravascular Lithotripsy (IVL) Technology in a Prospective, Multi-center, Single-arm Investigational Device Exemption (IDE) Study
Brief Title: FORWARD PAD IDE Study With the Shockwave Javelin IVL Catheter
Acronym: FORWARD PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 67398
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Arterial Disease
Keywords: Intravascular Lithotripsy
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- JAVELIN Study Catheter (Experimental): The JAVELIN catheter will be used to treat subjects with moderate to severely calcified peripheral artery disease (PAD) with target lesion located in a native, de novo superficial femoral, popliteal or infrapopliteal artery.
  Interventions: Device: Intravascular Lithotripsy

INTERVENTIONS:
Device: Intravascular Lithotripsy — The Shockwave Medical IVL System is intended for lithotripsy-enhanced treatment of lesions, including calcified lesions, to increase luminal diameter, allowing for further treatment (e.g. post-dilatation) in the peripheral arterial vasculature. Not for use in the coronary or cerebral vasculature.

SUMMARY:
The FORWARD PAD IDE Study is a prospective, multi-center, single-arm investigational device exemption study, conducted to assess the safety and effectiveness of the Shockwave Medical Mini S Peripheral IVL System for the treatment of heavily calcified, stenotic peripheral arteries.

ELIGIBILITY:
General Inclusion Criteria

1. Age of subject is ≥ 18 years.
2. Subject is able and willing to comply with all assessments in the study.
3. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate, and has signed the approved consent form.
4. Estimated life expectancy > 1 year.
5. Rutherford Clinical Category 2, 3, 4 or 5 of the target limb(s).

   Angiographic Inclusion Criteria
6. One or two target lesion(s) located in a native de novo superficial femoral, popliteal or infrapopliteal artery (above the ankle joint), in one or both limbs.
7. Target lesion reference vessel diameter (RVD) between 2.0 mm and 7.0 mm by investigator visual estimate.
8. Target lesion stenosis ≥70% (for vessels below the knee defined as P3 to the ankle joint) or ≥90% (for vessels above the knee) by investigator visual estimate.
9. Target lesion length is ≤150 mm by investigator visual estimate. Target lesion can be all or part of the 150 mm treated zone.
10. Calcification is at least moderate defined as presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending > 50% the length of the lesion if lesion is ≥50mm in length; or extending for minimum of 20mm if lesion is <50mm in length.

General Exclusion Criteria

1. Rutherford Clinical Category 0, 1 and 6 (target limb).
2. History of endovascular or surgical procedure on the target limb within the last 30 days or planned within 30 days of the index procedure, with the exception of toe amputation. Note: inflow treatment of non-target lesions is allowed providing successful treatment.
3. Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
4. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
5. Subject has known allergy to urethane, nylon, or silicone.
6. Myocardial infarction within 60 days prior to enrollment.
7. History of stroke within 60 days prior to enrollment.
8. Subject has acute or chronic renal disease with eGFR <30 ml/min/1.73 m2 (using CKD-EPI formula), unless on renal replacement therapy.
9. Subject is pregnant or nursing.
10. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
11. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
12. Covid-19 diagnosis within 30 days.
13. Planned use of cutting/scoring balloons, re-entry or atherectomy devices in target lesion(s) during the index procedure.
14. Planned major amputation of target limb.
15. Acute limb ischemia.
16. Occlusion of all the inframalleolar outflow arteries/vessels (i.e., desert foot).
17. Subject already enrolled into this study.

    Angiographic Exclusion Criteria
18. Failure to successfully treat clinically significant inflow lesions in the ipsilateral iliac, femoral, or popliteal arteries, defined as ≤30% residual stenosis with no serious angiographic complications (e.g. embolism).
19. Failure to successfully treat significant non-target infra-popliteal lesions, if treated prior to treatment of target lesion(s). Successful treatment is defined as obtaining ≤50% residual stenosis with no serious angiographic complications (e.g., embolism).
20. Target lesion includes in-stent restenosis.
21. Evidence of aneurysm or thrombus in target vessel.
22. No calcium or mild calcium in the target lesion.
23. Target lesion within native or synthetic vessel grafts.
24. Failure to successfully cross the guidewire across the target lesion; successful crossing defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2025-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Stanford Hospital and Clinics (SHC), Palo Alto, California
  - Advanced Heart and Vein Center, Thornton, Colorado
  - HCA Florida Blake Hospital, Bradenton, Florida
  - Tallahassee Memorial Healthcare, Inc., Tallahassee, Florida
  - UnityPoint Health Trinity Bettendorf Hospital, Bettendorf, Iowa
  - Cardiovascular Medicine PC, Davenport, Iowa
  - MedStar Montgomery Medical Center, Olney, Maryland
  - Southcoast Hospitals Group, New Bedford, Massachusetts
  - North Mississippi Medical Center, Tupelo, Mississippi
  - NYU Langone Health, New York, New York
  - Charlotte Radiology, Charlotte, North Carolina
  - The Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - Ascension St. John Jane Phillips Hosptial, Bartlesville, Oklahoma
  - Lankenau Institute for Medical Research, Bryn Mawr, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Heart Hospital Baylor, Plano, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Columbia St. Mary's, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | JAVELIN Study Catheter
Started | 55
30 Days Post-Procedure | 55
Completed | 0 (End of Study data not yet due for release)
Not Completed | 55

BASELINE CHARACTERISTICS:
Arm/Group | JAVELIN Study Catheter
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 48
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint - Major Adverse Events (MAE) at 30 Days
Description: Major Adverse Events (MAE) at 30 days defined as a composite of:
  * Cardiovascular death
  * Clinically-Driven Target Lesion Revascularization (CD-TLR)
  * Unplanned Target Limb Major Amputation (Above the Ankle)
Time Frame: 30 Days
Measure: Number; unit: participants
Arm/Group | JAVELIN Study Catheter
Number analyzed (Participants) | 55
participants
  Major Adverse Events | 0
  Cardiovascular Death | 0
  Clinically-Driven Target Lesion Revascularization (CD-TLR) | 0
  Unplanned Target Limb Major Amputation (Above the Ankle) | 0

2. Primary Outcome: Primary Effectiveness Endpoint - Technical Success
Description: Technical Success defined as final residual stenosis ≤50% without flow-limiting dissection (≥ Grade D) of the target lesion as assessed by angiographic core lab.
Time Frame: Peri-Procedural, immediately after all therapy of the target lesion was completed.
Population: Analysis was performed at the lesion level, where 55 subjects had 63 target lesions with evaluable data.
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | JAVELIN Study Catheter
Number analyzed (Participants) | 55
Number analyzed (Lesions) | 63
Lesions
  Technical Success | 62
  Freedom from Any Serious Flow-Limiting Dissection (D-F) | 62
  Residual Stenosis Less Than or Equal to 50% | 63

3. Secondary Outcome: Serious Angiographic Complications
Description: Defined as flow-limiting dissection (≥ Grade D), perforation, distal embolization, or acute vessel closure as assessed by the angiographic core laboratory
Time Frame: Peri-Procedural
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | JAVELIN Study Catheter
Number analyzed (Participants) | 55
Number analyzed (Lesions) | 63
Lesions | 1

4. Secondary Outcome: IVL Technical Success (Post- Dilatation)
Description: Defined as post-dilatation residual stenosis ≤50% without flow-limiting dissection (≥ Grade D) of the target lesion, as assessed by angiographic core laboratory (measured immediately following mandatory post-dilatation).
Time Frame: Peri-Procedural
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | JAVELIN Study Catheter
Number analyzed (Participants) | 55
Number analyzed (lesions) | 62
lesions
  IVL Technical Success (Post-dilatation) | 57
  Freedom from Any Serious Flow-Limiting Dissection (D-F) | 59
  Residual Stenosis ≤ 50% | 60

5. Secondary Outcome: IVL Device Success
Description: Defined as the ability to deliver, advance across the target lesion, pressurize, pulse, flush, and retrieve the Javelin IVL Catheter.
Time Frame: Peri-Procedural
Measure: Number; unit: Javelin Devices
Units Other Than Participants: Javelin Devices
Arm/Group | JAVELIN Study Catheter
Number analyzed (Participants) | 55
Number analyzed (Javelin Devices) | 71
Javelin Devices | 66

6. Secondary Outcome: Technical Success (Final)
Description: Defined as final residual stenosis of ≤30% without flow-limiting dissection (≥ Grade D) of the target lesion by angiographic core laboratory
Time Frame: Peri-Procedural
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | JAVELIN Study Catheter
Number analyzed (Participants) | 55
Number analyzed (Lesions) | 63
Lesions
  IVL Technical Success (Final) | 52
  Freedom from Any Serious Flow-Limiting Dissection (D-F) | 62
  Residual Stenosis ≤ 30% | 53

7. Secondary Outcome: MAEs at 6-months Post Procedure
Description: Major Adverse Events (MAEs) at 6 months defined as a composite of:
  * Cardiovascular Death
  * Clinically-driven Target Lesion Revascularization
  * Unplanned Target Limb Amputation (Above the Ankle)
Time Frame: 6 Months Post-Procedure
Reporting Status: Not Posted, anticipated posting 2025-11

8. Secondary Outcome: MAEs at 12-months Post Procedure
Description: Major Adverse Events (MAEs) at 12 months defined as a composite of:
  * Cardiovascular Death
  * Clinically-driven Target Lesion Revascularization
  * Unplanned Target Limb Amputation (Above the Ankle)
Time Frame: 12 Months Post-Procedure
Reporting Status: Not Posted, anticipated posting 2025-11

9. Secondary Outcome: Primary Patency at 12-Months
Description: * Above the knee lesions: freedom from ≥50% restenosis as determined by Duplex Ultrasound (DUS) and freedom from Clinically-Driven Target Lesion Revascularization (CD-TLR)
  * Below the knee lesions: freedom from both total occlusion (100% diameter stenosis by DUS) in all of the target lesions in a flow pathway, as well as a CD-TLR
Time Frame: 12-Months Post Procedure
Reporting Status: Not Posted, anticipated posting 2025-11

ADVERSE EVENTS:
Time Frame: 30-Days post-procedure.
Arm/Group | JAVELIN Study Catheter
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 10/55
Other Adverse Events (participants affected / at risk) | 20/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JAVELIN Study Catheter (N=55)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 2 (2)
Tendon Injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Foot amputation (Surgical and medical procedures) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JAVELIN Study Catheter (N=55)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (4)
Vascular procedure complication (Injury, poisoning and procedural complications) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT05858905/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT05858905/SAP_001.pdf